CLINICAL TRIAL: NCT02244450
Title: Evaluation of the Clinical Utility and Cost Effectiveness Ratio of Generalized Neonatal Screening for Severe Combined Immunodeficiencies (SCID) by Quantification of TRECs on Guthrie Cards
Brief Title: Generalized Neonatal Screening of Severe Combined Immunodeficiencies
Acronym: DEPISTREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RC14_0030
Record Dates: First submitted 2014-09-02; First posted 2014-09-19 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Severe Combined Immunodeficiency, Atypical
Keywords: Neonatal screening; severe combined immunodeficiency; T-cell Receptor Excision Circle
MeSH Terms: conditions — Severe combined immunodeficiency, atypical; Severe Combined Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screened patients (Experimental): SCID screening: more drops of blood are placed on a second Guthrie card when current screening (72 hours of life ) is performed after parents' information and consent. The card drawn for the protocol will follow the usual network except that the test for quantifying TRECs will be realized to determine the presence of SCID.
  Interventions: Biological: SCID screening
- Control group (No Intervention): SCID children diagnosed without screening by pediatricians local referents DIP

INTERVENTIONS:
Biological: SCID screening
  Arms: Screened patients

SUMMARY:
Severe combined Immunodeficiencies ( SCID ) are a group of inherited diseases of the immune system by characterised profound abnormalities of T cell development . Infants with SCID require prompt clinical response to Prevent life -threatening infection and studies show significantly improved survival in babies Diagnosed at birth as a result of previous family history . SCID follows criteria for population -based newborn screening since it is asymptomatic at birth and fatal within the first year of life, the confirmation of the disease is easy, there is a curative treatment , and it is known that early stem cell transplantation improves survival . Quantification of TRECs (T- cell receptor excision circles ) in DNA extracted from Guthrie samples is a sensitive screening test for Specific and SCID .

The investigators propose in this study to perform a neonatal screening of SCID , in a population of 200,000 babies over a period of two years .

The investigators propose to study the clinical utility and cost effectiveness ratio, and SCID screening to demonstrate that could result in a broad benefit to Individuals detected , making screening relatively cost-effective in spite of the low incidence of the disease .

DETAILED DESCRIPTION:
The project proposes to study the feasibility and cost-effectiveness ratio ( time management and life expectancy to 10 years) of generalized neonatal screening for SCID children by offering this screening to 200 000 children (100 000 children per year) over the entire territory. Prospective control group consists of children diagnosed with SCID out of 700,000 annual births who do not benefit from screening.

The protocol will be leant against the existing newborn screening , that is to say two more drops of blood are placed on a second Guthrie card when current screening (72 hours of life ) is performed after parents' information and consent. Eleven newborn screening regional associations will be involved with the inclusion of children in about 50 maternity hospitals. The card drawn for the protocol will follow the usual network except that the test for quantifying TRECs will be realized in two laboratories instead of eleven laboratories assigned to RA . Investigative Regional Associations (RAs) represent nearly 600,000 births / year and the amount of 200,000 children will be achieved in two years (duration of inclusion) . All children born in the participating maternity may be included if they meet the inclusion criteria. The result of the screening test for SCID will be available within 21 days after birth, provided that there is no need to request a new sample.

At each of eleven RA is associated a pediatrician referent for immune deficiencies, member of the french reference center (CEREDIH) and who will be responsible to call the parents, offer them a consultation and further exploration if the result of screening is assumed positive.

Analysis of cards from 200,000 children will give the following information:

* Number of children with a presumptive positive screening , requiring a call by the referent pediatrician, consultation and exploration of lymphocyte subpopulations
* Number of children with a negative screening
* Number of children with an inconclusive screening (lack of TRECs and lack of amplification of the reference gene) and requiring a new card,

A micro- costing study will be conducted to assess the cost of testing .

This group of 200,000 children is the experimental group to assess the cost of screening , acceptability by parents (participation rate), the recall rate for abnormal or inconclusive result, the rate of follow-up time for results , the incidence of disease . It will also allow to calculate the specificity of the method .

At the end of the inclusions, the vital status at 18 months with cause of death will be sought for the 200 000 children included , with the CESP ( Centre de Recherche en Epidemiologie et Santé des Populations) via RNIPP (Répertoire National d'Identification des Personnes Physiques) and CepiDc ( Centre d'Epidémiologie sur les causes médicales de décès) . This will establish whether there are SCID in this population which were not detected at birth. Furthermore, the investigators include in the study SCID children diagnosed without screening by pediatricians local referents DIP (including Necker main transplant center) . This will enable to approach the sensitivity of the method . All these data allow the calculation of the predictive values of the test.

In this experimental group will be isolated a group of individuals who screened positive and diagnosed as true SCID . Clinical data for these patients will be collected in an electronic CRF ( CRF ) by the pediatrician referral protocol (Dr Thomas C ) , including:

* The dates and results of explorations : lymphocyte subpopulations , blood count, determination of immunoglobulin levels
* The diagnosis made with identification of the genetic defect
* The date of care before curative treatment ( protected area isolation , anti -infective drugs )
* , Bacterial , fungal anti -viral treatments , and other
* The date of transplant, type of transplant or other treatment ... ...

ELIGIBILITY:
Inclusion Criteria:

* Screening Group: Newborn on day 3 of birth (premature and non premature)
* Control group: Patients diagnosed with SCID without screening at participating centers

Exclusion Criteria:

* Lack of parental consent
* Children whose parents are adults under guardianship,
* Children without health insurance, for the screening group:
* The early exit of the child from the maternity hospital

Ages: 3 Days to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190539 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
cost / efficiency ratio of the implementation of the generalized neonatal screening of SCID at birth | 18 months
  Efficacy endpoint: number of children receiving early therapeutic suitable for curative ( transplant, enzyme treatment or gene therapy)

SECONDARY OUTCOMES:
Cost / efficiency ratio of the implementation of the generalized neonatal screening of SCID at birth | 10 years
  Efficacy endpoint: life expectancy of children modeled from the results of the study and data from the literature
The cost of care during the first 18 months of life per child enjoying an early curative treatment in the first 4 months of life. | 18 months
  Costs of care will be estimated during the first 18 months of life of the child.
Length of hospitalization of children with SCID in the first 18 months of life | 18 months
number of avoided deaths | 18 months
number of detected SCID patients | 18 months
number of patients detected with other T lymphopenia (SCID variants , DiGeorge , severe T lymphopenia non SCID ... ) | 18 months
number of false negative and false positive results | 18 months
  False negative results : patients from the control group diagnosed with SCID without screening who would have a negative screening or patients from the screening group died from a SCID and with a negative screening False positive: patients from the screening group with a positive screening but without SCID

CONTACTS AND LOCATIONS:
Overall Officials: Caroline THOMAS, MD, Principal Investigator — Nantes University Hospital; Marie AUDRAIN, MD, Study Director — Nantes University Hospital; Sophie MIRALLIE, Principal Investigator — Nantes University Hospital
Locations (50):
- France (50):
  - Angers Private Hospital Clinique de l'Anjou, Angers
  - Angers University Hospital, Angers
  - Argenteuil Hospital, Argenteuil
  - Aulnay-sous-Bois Hospital CHI Robert Ballanger, Aulnay-sous-Bois
  - Bordeaux Maison de Santé Protestante Bordeaux Bagatelle, Bordeaux
  - Bordeaux Private Hospital Polyclinique Bordeuax Nord Aquitaine, Bordeaux
  - Bordeaux University Hospital, Bordeaux
  - Corbeil Essonnes Hospital Sud Francilien, Corbeil-Essonnes
  - Créteil Hospital, Créteil
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital, Grenoble
  - Le Blanc Mesnil Private Hospital, Le Blanc-Mesnil
  - Lens Hospital, Lens
  - Libourne Maternity Hospital, Libourne
  - Lille University Hospital, Lille
  - Lormont Maternity Hospital Rive Droite, Lormont
  - Lyon Maternity Hospital, Lyon
  - Lyon University Hospital, Lyon
  - Marseille Saint-Joseph Hospital, Marseille
  - Marseille University Hospital La Conception, Marseille
  - Marseille University Hospital Nord, Marseille
  - Marseille University Hospital, Marseille
  - Meaux Hospital, Meaux
  - Montreuil Hospital CHI André Grégroie, Montreuil
  - Nantes University Hospital, Nantes
  - Nantes Private Hospital Clinique Jules Verne, Nantes
  - Paris Hospital Saint-Joseph, Paris
  - Paris Necker University Hospital, Paris
  - Paris University Hospital Armand-Trousseau, Paris
  - Paris University Hospital Bichat, Paris
  - Paris University Hospital Bicêtre, Paris
  - Paris University Hospital Béclère, Paris
  - Paris University Hospital Jean Verdier, Paris
  - Paris University Hospital La Pitié Salpétrière, Paris
  - Paris University Hospital Louis Mourier, Paris
  - Paris University Hospital Necker, Paris
  - Poissy Hospital CHI Poissy-Saint-Germain, Poissy
  - Pontoise Hospital René Dubos, Pontoise
  - Rennes Private Hospital Clinique Mutualiste La Sagesse, Rennes
  - Rennes University Hospital, Rennes
  - Saint-Grégoire Private Hospital, Rennes
  - Roubaix Hospital, Roubaix
  - Saint-Herblain Private Hospital Polyclinique de l'Atlantique, Saint-Herblain
  - Saint-Mande Army Hospital Begin, Saint-Mandé
  - Saint-Martin-d'Hère Private Hospital Clinique Belledonne, Saint-Martin-d'Hères
  - Strasbourg Private Hospital Clinique Adassa, Strasbourg
  - Strasbourg University Hospital, Strasbourg
  - Toulouse Private Hospital Clinique Sarrus Teinturiers, Toulouse
  - Toulouse University Hospital P. DE VIGUIER, Toulouse
  - Toulouse University Hospital, Toulouse

REFERENCES:
- [Derived] Thomas C, Durand-Zaleski I, Frenkiel J, Mirallie S, Leger A, Cheillan D, Picard C, Mahlaoui N, Riche VP, Roussey M, Sebille V, Rabetrano H, Dert C, Fischer A, Audrain M. Clinical and economic aspects of newborn screening for severe combined immunodeficiency: DEPISTREC study results. Clin Immunol. 2019 May;202:33-39. doi: 10.1016/j.clim.2019.03.012. Epub 2019 Apr 1. PMID 30946917
- [Derived] Audrain MAP, Leger AJC, Hemont CAF, Mirallie SM, Cheillan D, Rimbert MGM, Le Thuaut AM, Sebille-Rivain VA, Prat A, Pinel EMQ, Divry E, Dert CGL, Fournier MAG, Thomas CJC. Newborn Screening for Severe Combined Immunodeficiency: Analytic and Clinical Performance of the T Cell Receptor Excision Circle Assay in France (DEPISTREC Study). J Clin Immunol. 2018 Oct;38(7):778-786. doi: 10.1007/s10875-018-0550-7. Epub 2018 Sep 24. PMID 30251145